CLINICAL TRIAL: NCT04602338
Title: Multimodality Imaging (Cardiovascular Magnetic Resonance Imaging, Echocardiography, and Nuclear Medicine Imaging) in the Screening, Diagnosis and Risk Stratification of Heart Failure With Preserved Ejection Fraction- a Multicenter Study.
Brief Title: Diagnosis and OutcoMes evaluAtIoN of Multicenter Patients With HFpEF Using Multimodality Imaging
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Anzhen Hospital (Other); China-Japan Friendship Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, Vice Director of Magnetic Resonance Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: DOMAIN-HFPEF
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure, Diastolic; Multicenter Study
Keywords: heart failure with preserved ejection fraction; cardiovascular magnetic resonance imaging; echocardiography; nuclear medicine imaging; early diagnosis; prognosis
MeSH Terms: conditions — Heart Failure, Diastolic; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples Without DNA — data of radiology imaging, clinical study and laboratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of Heart failure with preserved ejection fraction (HFpEF) in Heart failure patients increases rapidly. However, the current clinical awareness is insufficient, and the cardiac structural and functional injury are not well understood. It is difficult to recognize the subclinical changes of the cardiac in the early stage with conventional imaging techniques, and it is common to ignore the existence of the clinical alterations. This study aimed to investigate the cardiac features, early diagnosis and risk factors of HFpEF patients, based on the multi-modality (Magnetic resonance imaging- nuclear medicine imaging- echocardiography) imaging and multicenter study, combined with large data and artificial intelligence. This study will provide deep insights into the HFpEF in multicenter population.

DETAILED DESCRIPTION:
Heart Failure with Preserved Ejection Fraction (HFpEF) is a special subtype of Heart Failure (HF), and the incidence of HF cases is rising to 4.5 million every year, according to "Chinese cardiovascular disease report 2018" and "China Heart Failure and diagnostic guidelines 2018". In 2000, the incidence of patients with chronic Heart Failure is as high as 0.9%, and faces significantly increase with the increase of age. Moreover, HFpEF patients accounted for over 50% of heart failure, presenting normal left ventricular ejection fraction (LVEF), and nonspecific HF clinical performance. In addition, as a heterogenous disease, HFpEF is often associated with various comorbidities, including hypertension (~ 75%), diabetes (~ 40%), obesity (> 80%), aging (~ 75 years), renal dysfunction (25-50%), pulmonary hypertension (~ 50%), and other diseases. There is still much confusion about the pathophysiology of the disease, and no effective treatment was confirmed, therefore the diagnosis and treatment HFpEF has some challenges. With the increase of cardiovascular risk factors such as hypertension (morbidity: 23.2% in 2018), diabetes (morbidity:10.9% in 2018, treatment rate 32.2%) and the aging trend, the morbidity and mortality of HFpEF are still on the rise, posing a threat to the life quality of more and more patients. Early identification and intervention of HFpEF is an important method to reduce mortality and improve prognosis. Yet, many studies have explored the role of different biochemical and inflammatory markers in the diagnosis and prognosis assessment of HFpEF, limited for mixed indicators and low sensitivity.

Cardiac Magnetic Resonance imaging (CMR) is a non-invasive "one-stop" examination, including cardiac structure, function, tissue characteristics, blood perfusion examination. In particular, the emerging T1 mapping and Feature Tracking (FT) techniques enable the early and quantitive identification of cardiac dysfunction prior to abnormal LVEF. It has been found that the Extracellular Volume Fraction (ECV) based on T1 mapping and the myocardial strain parameters based on FT have the ability to diagnose and predict the prognosis of HFpEF patients. Echocardiography takes advantages in early identification of HFpEF patients and reveals the diastolic dysfunction. Nuclear medicine imaging shows priorities in blood perfusion and myocardial viability verification. Magnetic resonance imaging - echocardiography - nuclear medicine multimodal imaging complements and promotes each other, for example, molecular nuclear medicine imaging (recognition of metabolism), echocardiography (primary selection and determination of diastolic dysfunction), as well as the noninvasive high-resolution magnetic resonance and new emerging molecular imaging (identification of macroscopic, microscopic structure and function). The multimodel imaging overcomes the limits of single imaging method, greatly improves the accuracy of early diagnosis ability and diagnosis. However, large studies are based on single-center studies and meta analysis of small samples, and the comprehensive markers derived from multimodel study and multicenter study are lacked. Domestic relevant studies are in the initial stage.

To sum up, this study attempts to achieve early diagnosis and intervention of HFpEF and improve life quality of HFpEF patients through a multicenter, large sample cooperative study based on multimodel imaging (CMR imaging, echocardiography, nuclear medicine imaging). This study is expected to deepen the understanding of the pathogenesis and pathophysiological characteristic of HFpEF, providing a set of parameters based on multimodel imaging, hence assisting in early identification of cardiac structure and function change, early diagnosis of HFpEF and achieving risk stratification. In other way, the marker derived from this study may help target treatment of HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction (LVEF)≥50%；
* N-terminal pro-b type natriuretic peptide (NT-proBNP)>220pg/ml or b type natriuretic peptide (BNP) >80 pg/ml;
* symptoms and syndromes of heart failure;
* At least one criteria of cardiac structure (left ventricular hypertrophy, or left atrial enlargement) and function abnormalities (based on tissue doppler, color doppler).

Exclusion Criteria:

* Special types of cardiomyopathy, including hypertrophic cardiomyopathy, restricted cardiomyopathy, etc.
* Infarction, myocardial fibrosis caused by ischemic cardiomyopathy and acute coronary syndrome ;
* Severe arrhythmia;
* Severe primary cardiac valvular disease;
* Restrictive pericardial disease;
* Refuse to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study is a prospective, multicenter study with HFpEF patients, diagnosed based on 2016 and 2019 European Society of Cardiology (ESC) concensus. The inclusion criteria include left ventricular ejection fraction (LVEF)≥50%；N-terminal pro-b type natriuretic peptide (NT-proBNP)>220pg/ml or b type natriuretic peptide (BNP) >80 pg/ml; symptoms and syndromes of heart failure; and at least one criteria of cardiac structure (left ventricular hypertrophy, or left atrial enlargement) and function abnormalities. We exclude patients with special cardiomyopathy, ; Infarction, myocardial fibrosis caused by ischemic cardiomyopathyand acute coronary syndrome; Severe arrhythmia; Severe primary cardiac valvular disease; Restrictive pericardial disease; Refuse to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
All-cause Death | 1-8 year
  the incidence of all-cause death
Cardiovascular Death | 1-8 year
  the incidence of cadridovascular death
Hospitalization Due to Heart Failure | 1-8 year
  the incidence of Hospitalization Due to Heart Failure

SECONDARY OUTCOMES:
Implantable cardioverter-defibrillator Implantation | 1-8 year
  the incidence of Implantable cardioverter-defibrillator Implantation
Heart Transplantation | 1-8 year
  the incidence of Heart Transplantation
Pacemaker Implantation | 1-8 year
  the incidence of Pacemaker Implantation
Atrial fibrillation | 1-8 year
  the incidence of Atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Minjie Lu, PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Our study data is applicable to other researchers with permmsion.

REFERENCES:
- [Result] Tsao CW, Lyass A, Enserro D, Larson MG, Ho JE, Kizer JR, Gottdiener JS, Psaty BM, Vasan RS. Temporal Trends in the Incidence of and Mortality Associated With Heart Failure With Preserved and Reduced Ejection Fraction. JACC Heart Fail. 2018 Aug;6(8):678-685. doi: 10.1016/j.jchf.2018.03.006. Epub 2018 Jul 11. PMID 30007560
- [Result] Shah SJ, Kitzman DW, Borlaug BA, van Heerebeek L, Zile MR, Kass DA, Paulus WJ. Phenotype-Specific Treatment of Heart Failure With Preserved Ejection Fraction: A Multiorgan Roadmap. Circulation. 2016 Jul 5;134(1):73-90. doi: 10.1161/CIRCULATIONAHA.116.021884. PMID 27358439
- [Result] Altara R, Giordano M, Norden ES, Cataliotti A, Kurdi M, Bajestani SN, Booz GW. Targeting Obesity and Diabetes to Treat Heart Failure with Preserved Ejection Fraction. Front Endocrinol (Lausanne). 2017 Jul 17;8:160. doi: 10.3389/fendo.2017.00160. eCollection 2017. PMID 28769873
- [Result] De Keulenaer GW, Brutsaert DL. Systolic and diastolic heart failure: different phenotypes of the same disease? Eur J Heart Fail. 2007 Feb;9(2):136-43. doi: 10.1016/j.ejheart.2006.05.014. Epub 2006 Aug 1. PMID 16884955
- [Result] Campbell RT, McMurray JJ. Comorbidities and differential diagnosis in heart failure with preserved ejection fraction. Heart Fail Clin. 2014 Jul;10(3):481-501. doi: 10.1016/j.hfc.2014.04.009. PMID 24975911
- [Result] Guazzi M. Pulmonary hypertension in heart failure preserved ejection fraction: prevalence, pathophysiology, and clinical perspectives. Circ Heart Fail. 2014 Mar 1;7(2):367-77. doi: 10.1161/CIRCHEARTFAILURE.113.000823. No abstract available. PMID 24643889
- [Result] Simmonds SJ, Cuijpers I, Heymans S, Jones EAV. Cellular and Molecular Differences between HFpEF and HFrEF: A Step Ahead in an Improved Pathological Understanding. Cells. 2020 Jan 18;9(1):242. doi: 10.3390/cells9010242. PMID 31963679
- [Result] Loai S, Cheng HM. Heart failure with preserved ejection fraction: the missing pieces in diagnostic imaging. Heart Fail Rev. 2020 Mar;25(2):305-319. doi: 10.1007/s10741-019-09836-8. PMID 31364028
- [Result] Marwick TH, Shah SJ, Thomas JD. Myocardial Strain in the Assessment of Patients With Heart Failure: A Review. JAMA Cardiol. 2019 Mar 1;4(3):287-294. doi: 10.1001/jamacardio.2019.0052. PMID 30810702
- [Result] Su MY, Lin LY, Tseng YH, Chang CC, Wu CK, Lin JL, Tseng WY. CMR-verified diffuse myocardial fibrosis is associated with diastolic dysfunction in HFpEF. JACC Cardiovasc Imaging. 2014 Oct;7(10):991-7. doi: 10.1016/j.jcmg.2014.04.022. Epub 2014 Sep 17. PMID 25240451
- [Result] Harinstein ME, Soman P. Radionuclide Imaging Applications in Cardiomyopathies and Heart Failure. Curr Cardiol Rep. 2016 Mar;18(3):23. doi: 10.1007/s11886-016-0699-8. PMID 26841785
- [Result] Recommendations for Cardiac Chamber Quantification by Echocardiography in Adults: An Update from the American Society of Echocardiography and the European Association of, Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2016 Apr;17(4):412. doi: 10.1093/ehjci/jew041. Epub 2016 Mar 15. No abstract available. PMID 26983884
- [Result] Schnelle M, Catibog N, Zhang M, Nabeebaccus AA, Anderson G, Richards DA, Sawyer G, Zhang X, Toischer K, Hasenfuss G, Monaghan MJ, Shah AM. Echocardiographic evaluation of diastolic function in mouse models of heart disease. J Mol Cell Cardiol. 2018 Jan;114:20-28. doi: 10.1016/j.yjmcc.2017.10.006. Epub 2017 Oct 19. PMID 29055654